CLINICAL TRIAL: NCT06748287
Title: A Clinical Comparison of FDA-Cleared Photobiomodulation Devices for the Treatment of Alopecia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DERM-2017-25394
Record Dates: First submitted 2024-04-26; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- iGrow Hair Growth System (Experimental): male or female subjects ages 21-85 with alopecia randomized to use iGrow Hair Growth System photobiomodulation device.
  Interventions: Device: iGrow Hair Growth System
- Capillus352 (Active Comparator): male or female subjects ages 21-85 with alopecia randomized to use Capillus352 photobiomodulation device.
  Interventions: Device: Capillus352
- HairMax Ultima 12 Lasercomb (Experimental): male or female subjects ages 21-85 with alopecia randomized to use HairMax Ultima 12 Lasercomb photobiomodulation device.
  Interventions: Device: HairMax Ultima 12 Lasercomb
- HairMax Laserband 82 (Experimental): male or female subjects ages 21-85 with alopecia randomized to use HairMax Laserband 82 photobiomodulation device.
  Interventions: Device: HairMax Laserband 82

INTERVENTIONS:
Device: iGrow Hair Growth System — has a helmet-design and headphones to allow for hands-free use and music listening capabilities. Treatment is 25 minutes every other day. three to four times per week for 4 months.
  Arms: iGrow Hair Growth System
Device: Capillus352 — has a similar design to a salon hair dryer which hovers over the head to allow for hand-free use. Treatment is 12 minutes, three times per week for 4 months.
  Arms: Capillus352
Device: HairMax Ultima 12 Lasercomb — is comb-like device with hair-parting teeth to aid in delivery of light therapy directly to the scalp. Treatment is 8 minutes three times per week for 4 months.
  Arms: HairMax Ultima 12 Lasercomb
Device: HairMax Laserband 82 — is headband design device which has unique hair-parting teeth to aid in delivery of light therapy directly to the scalp. Treatment is 90-second treatments three times per week for 4 months.
  Arms: HairMax Laserband 82

SUMMARY:
Photobiomodulation is a form of non-ionizing light therapy has been shown to stimulate cellular processes and reduce inflammation as well as improve pain and wound healing. Photobiomodulation has also been found to enhance fibroblast growth factor production. A challenge in clinic is to answer the patients' questions regarding which FDA-cleared device is the best to purchase. Therefore, this study was designed to gain experience with the use of the following devices and to clinically evaluate their efficacy: iGrow Hair Growth System, Capillus352, Hair Max Ultima 12 LaserComb, and HairMax Laserband 82. The purpose of this pilot research study is to clinically compare and evaluate FDA-cleared photobiomodulation devices after four months of treatment and one-month follow-up in subjects with alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 21-85 years old with alopecia.
* Prospective subjects must be in good general health.
* Female subjects who are premenopausal and of childbearing capacity must use oral contraceptive tablets, implanted contraceptive hormones, or Depo-Provera® contraceptive injections as birth control for the duration of the study.
* If prospective subjects are on hormone-containing medication, they must be on stable dose for past 6 months.
* Willing to abstain from use of over-the-counter hair products such as topical Minoxidil (Rogaine ® ) and prescription hair products.
* Willing to use DHS zinc shampoo and conditioner for the duration of the study.
* Willing to avoid using any hair styling products directly on the scalp.
* Subjects must be capable of giving informed consent.
* Willing to adhere to protocol, including scalp examinations, questionnaires, and photography.
* Willing to adhere to treatment protocol and frequency used for FDA clearance.
* Willing to retain the same hair style and color throughout the duration of the study.
* Willing to shampoo/clean scalp at least 3 times per week.

Exclusion Criteria:

* Immunosuppressed patients (history of transplantation, cancer, chemotherapy, splenectomy, or HIV)
* Application of topical immunomodulatory or immunosuppressive agent in the preceding 6 weeks.
* Systemic administration of corticosteroid or other systemic treatment (i.e., prednisone) that has immunomodulatory or other immunosuppressive mechanisms of action, in the preceding 3 months or planned usage throughout the study.
* Clinical evidence of secondary skin infection (i.e., folliculitis).
* Other scalp conditions (i.e., seborrheic dermatitis or dissecting cellulitis) that might interfere with evaluations during the study.
* Investigational medications within the past 30 days.
* Female prospective subject is pregnant, nursing, planning a pregnancy, or less than six months postpartum.
* Severe allergies manifested by a history of anaphylaxis, or history or presence of multiple severe allergies.
* Use of photobiomodulating device, such as those in this study, within the past 4 weeks
* Initiation or change in dose/application of topical minoxidil within the past 6 weeks.
* Finasteride or dutasteride within the last 3 months.
* Spironolactone within the past 3 months.
* Vitamin supplementation (i.e. selenium, or biotin) in excess of daily recommendation per manufacturer.
* Lesions in the treated area suspicious for malignancy, or prior skin cancer.
* Radiation or chemotherapy to the scalp.
* Use of topical or oral ketoconazole in the past 4 weeks.
* Hair transplant procedure within the past 6 months or throughout the duration of the study.
* History of microneedling procedure performed on scalp.
* Changes in hair style while enrolled in the study.
* Current weave, or plans to get a weave while enrolled in the study.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment Score (IGA score) | baseline to 5 months
  Units on a scale. Standardized rating system used in research to assess various dermatologic conditions, including hair loss (-3-+3). It involves visual examination by trained board-certified dermatologists to evaluate specific criteria assessing the overall severity of hair loss.
Savin score | baseline to 5 months
  Units on a scale. Classification systems for female pattern hair loss (I-1-III) severity, assessed during monthly examinations.
Ludwig score | baseline to 5 months
  Units on a scale. Classification system for female pattern hair loss (I-III) severity, assessed during monthly examinations.
Hamilton-Norwood score | Baseline to 5 months
  Units on a scale. Classification systems for male pattern hair loss (I-VII) severity, assessed during monthly examinations.
Dermatologist Evaluation of Scalp Health (Scale) | Baseline to 5 months
  Scalp health, specifically scale, is evaluated and marked as "absent", "mild", or "moderate" by a board-certified dermatologist during monthly examinations.
Dermatologist Evaluation of Scalp Health (Erythema) | Baseline to 5 months
  Dermatologist Evaluation of Scalp Health (Erythema) Description: Scalp health, specifically erythema, is evaluated and marked as "absent", "mild", or "moderate" by a board-certified dermatologist during monthly examinations.
Dermatologist Evaluation of Scalp Health (Folliculitis) | Baseline to 5 months
  Scalp health, specifically folliculitis, is evaluated and marked as "absent", "mild", or "moderate" by a board-certified dermatologist during monthly examinations.
Hair Growth Assessment (HGA) | Baseline to 5 months
  Units on a scale. A scale used to describe scalp hair growth progress compared to baseline photos. Change is quantified on a scale of -3 to 3.
Hair Growth Index (HGI) | Baseline to 5 months
  Units on a scale. Hair growth is evaluated using three self-assessment questions on a scale of -3 to 3.
Hair Growth Satisfaction Surveys (HGSS) | Baseline to 5 months
  Units on a scale. Participant satisfaction with hair appearance/growth compared to baseline across five questions on a scale of -3 to 3.
Subject Scalp Health Assessment (SSHA) | Baseline to 5 months
  Units on a scale. Self-assessment of scalp health and hair condition through multiple questions measured on a scale of -2 to 2 during monthly exams.

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States